CLINICAL TRIAL: NCT05183633
Title: A Pilot Study to Assess the Association Between Human Bioimpedance Measurements and Clinical Urodynamic Procedures
Status: Terminated | Type: Observational
Why Stopped: Was not able not determine a meaningful bioimpedance measurement that could be correlated to bladder fullness over time.
Sponsor: Curbell Medical Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HRP-503
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Patients Susceptible to Falls

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One single trial

SUMMARY:
A Pilot Study to Assess the Association between Human Bioimpedance Measurements and Clinical Urodynamic Procedures

DETAILED DESCRIPTION:
The purpose of the study is to assess how well Curbell's Bladder Sensor device measuring bioimpedance correlates to urodynamic studies and the reported sensation subjects feel when reporting bladder fullness and their urge to urinate.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have been previously scheduled for a Urodynamic Study

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have been previously scheduled for a urodynamic study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Correlation of Urge to Urinate to Bioimpedance. Our clinical trial is an attempt to determine the correlation of bioimpedance measurements versus bladder pressure (fullness) taken at the same time during a normally scheduled urodynamic study. | Bioimpedance measurements are taken in real time simultaneously with urodynamic pressure measurements. Therefore, the time frame is "zero." Each measurement characterizes actual bioimpedance at that point in time.
  Our primary outcome is determining the correlation strength between the bladder's pressure measurements (acquired during a standard urodynamic study) and bioimpedance measurements. That is, we are trying to find if bladder bioimpedance is correlated to bladder fullness, where pressure is the clinically-accepted measurement of bladder fullness in a urodynamic study.

CONTACTS AND LOCATIONS:
Locations (1):
- Western New York Urology Associates, Cheektowaga, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided